CLINICAL TRIAL: NCT01358656
Title: Comparison of the Anterior Cruciate Ligament Reconstruction Using Single Bundle and Double Bundle Techniques: Prospective Clinical Study
Brief Title: Anterior Cruciate Ligament Reconstruction Using Single Bundle and Double Bundle Techniques
Acronym: KR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vita Care (Other)
Responsible Party: Vita Care, Vita Care
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KR
Record Dates: First submitted 2011-05-19; First posted 2011-05-24 (Estimated); Last update posted 2011-05-24 (Estimated); Status verified 2011-05

CONDITIONS: Anterior Cruciate Ligament Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single Bundle Reconstruction (Active Comparator): Subjects will undergo single bundle acl reconstruction
  Interventions: Procedure: Single bundle anterior cruciate ligament reconstruction
- Double bundle reconstruction (Active Comparator): Subjects will undergo double bundle acl reconstruction
  Interventions: Procedure: Double bundle anterior cruciate ligament reconstruction

INTERVENTIONS:
Procedure: Single bundle anterior cruciate ligament reconstruction — The surgical technique includes ACL reconstruction with graft of two autologous tendons - the semitendinous and gracilis - fixed in one tibial tunnel and one femoral tunnel. Once the graft is obtained, the arthroscopy-assisted ACL reconstruction is performed using anterolateral, anteromedial and accessory anteromedial portals. The first tunnel to be built is femoral tunnel, through a Smith & Nephew femoral guide inserted into the anteromedial portal in the 10:30 h position for the right knee and 1:30 h position for the left knee, with the knee at 120° of flexion. The next tunnel is tibial tunnel. The tunnel has its point of entry anterior to the fibers of the superficial medial collateral ligament, and the tibial guide must be adjusted at 45 degrees. The new ligament is fixed onto the tibia and femur with a biodegradable interference screw.
  Arms: Single Bundle Reconstruction
Procedure: Double bundle anterior cruciate ligament reconstruction — The ACL reconstruction is performed with graft of two autologous tendons -the semitendinous and gracilis- fixed in two tibial tunnels and two femoral tunnels. The first tunnel to be built is the anteromedial (AM) femoral tunnel, through femoral guide inserted into the AM portal in the 10:30 h position for the right knee and 1:30 h position for the left knee, with the knee at 120° of flexion. Then we drill the PL femoral tunnel in its anatomical position from the accessory AM portal, with the knee at 120° of flexion. The next tunnels are the PM and AM tunnels. The PL tunnel has its point of entry anterior to the fibers of the superficial medial collateral ligament, and the tibial guide must be adjusted at 45º. The AM tunnel has its point of entry more lateral, and a bone bridge of at least one cm must be left between the tunnels, and the tibial guide adjusted at 55º. Both bundles must be fixed onto the tibia and femur with a biodegradable interference screw.
  Arms: Double bundle reconstruction

SUMMARY:
Anterior Cruciate Ligament (ACL) reconstruction surgery has greatly advanced over the last 20 years. However, data in the literature reveal that approximately 15-25% of patients undergoing surgery still do not present optimal outcomes, which suggests that there is room for improvement of the procedure. A possible explanation for this fact is that most ACL reconstructions consider only one of the functional bundles of the ligament. Our hypothesis is that the ACL reconstruction with the double-bundle technique will be effective in reducing the patients' rotation of the knee joint for high-demanding tasks compared to the patients who had ACL reconstruction with the single-bundle technique.

DETAILED DESCRIPTION:
The aim of this study is to compare the ACL reconstruction with only one bundle (one tunnel in the tibia and femur) with the procedure to reconstruct the the ACL with two bundles with 2 tunnels in the tibia and 2 in the femur (considered closest to the normal anatomy of of the ACL), both in terms of objective and subjective results.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female.
2. Body mass index (BMI), which corresponds to the ratio between weight in kilograms (pounds) and height in m2 (square meters) between 18.5 and 24.99.
3. Anterior instability alone or associated with chondral lesions of up to 1cm or associated with meniscal injuries that do not alter the postoperative rehabilitation.
4. Magnetic resonance imaging (MRI) confirming the ACL injury.
5. Aged between 20 and 45 years.
6. Not having asymmetric varus alignment, greater than or equal to 5 degrees (to eliminate cases with indication for osteotomy of the tibia), using panoramic radiographic comparison of the lower limbs in standing position.
7. Absence of associated ligament instabilities (medial, lateral or posterior).
8. No previous surgery on the affected knee.

Exclusion Criteria:

1. New post-surgical trauma after 12 months.
2. Interruption of treatment / follow-up.
3. Postoperative infection.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-07 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Isokinetic testing | 2 years
  Tests the muscle power and endurance
Subjective and Objective IKDC Scores | 2 years
  The subject will answer the subjective IKDC score and the investigator will complete the objective IKDC score
Kinematic evaluation | 2 years
  The subjects will perform 3 tasks. Walking with no change of direction. Walking with change of direction: walk straight until one foot will touch the force platform and at that moment the subject must change their direction of motion and make a 90° angle with respect to the original trajectory by rotating the body to the side of the foot that will touch the platform. Landing with change of direction: step down 4 steps of a stair as they touch the force platform in the ground, they change the direction of their motion so that the new trajectory will make a 90° angle with the former direction.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Vita, São Paulo, São Paulo, Brazil